CLINICAL TRIAL: NCT00029276
Title: Transcranial Magnetic Stimulation For Treatment Of Depression In Parkinson's Disease
Brief Title: Magnetic Stimulation for Parkinson Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01AT000610-01 (NIH)
Record Dates: First submitted 2002-01-09; First posted 2002-01-10 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Parkinson's Disease; Depression
Keywords: Parkinson's; Depression; Magnetic Stimulation
MeSH Terms: conditions — Parkinson Disease; Depression

INTERVENTIONS:
Procedure: Prefrontal transcranial magnetic brain stimulation

SUMMARY:
During transcranial magnetic stimulation (TMS), a magnetic coil is placed on the front part of the head. Electric current passes through the coil in brief pulses. Magnetism from the current produces a separate, small electric current inside the brain, which activates brain cells below the coil. This treatment may result in decreased depression and improved Parkinson's disease symptoms.

DETAILED DESCRIPTION:
The major aim of this study is to carry out a sequential Phase I trial of prefrontal transcranial magnetic brain stimulation (TMS) and electroconvulsive therapy (ECT) in patients with Parkinson's disease (PD) and severe depression. Depression complicates PD in up to 50% of cases, leading to further deterioration of motor performance and quality of life; but antidepressant medication fails or produces intolerable side effects in 25-30% of patients. Case reports and uncontrolled trials suggest that ECT is effective in ameliorating simultaneously the mood and motor symptoms of PD. Only a few small studies of ECT in PD have been prospective or randomized, the assessment protocols have been limited, and the results have been variable. TMS is a new, promising, alternative treatment for refractory depression, which appears to be easier and safer than ECT. Requiring no hospitalization, anesthesia, or recovery time, TMS is now being investigated as an alternative therapy for mood disorders. TMS has not been studied in depressed patients with PD or in other serious central nervous system diseases.

This study extends our past and present research in PD, depression, ECT, and TMS. We will comprehensively evaluate the effects of left prefrontal TMS on mood, motor, and neuropsychological function, together with quality of life indices in depressed PD patients. All patients will initially receive treatment with TMS. Those who fail to benefit will proceed to ECT. Comprehensive evaluation will be continued for another eight weeks in both the TMS-only and ECT groups. The key issues addressed by these studies include: (1) the potential benefit of TMS on mood and movement in depressed PD patients, and (2) the tightness of the association between mood and motor function after TMS and ECT. Overall, these studies will provide important preliminary data on the relationships among mood, cognitive and motor function in PD, and their influence on quality of life. The results will help in directing future applications of TMS as an alternative therapy for brain disorders, and will further elucidate the relative benefits of both TMS and ECT in depressed PD patients. A positive effect from TMS should be an impetus towards randomized, placebo-controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of idiopathic Parkinson's Disease and meet DSM-IV criteria for Major Depressive Episode, severe, with or without psychotic features, or for Mood Disorder secondary to PD with major depression-like episode.
* Have demonstrated an inadequate clinical response to at least one antidepressant medication in adequate dosage for at least six weeks, or an adverse event requiring discontinuation.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2000-08; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Charles Epstein, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States